CLINICAL TRIAL: NCT04064567
Title: Linking High-Risk Jail Detainees to HIV Pre-Exposure Prophylaxis: PrEP-LINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 239250
Record Dates: First submitted 2019-08-14; First posted 2019-08-22 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: HIV/AIDS; Pre-exposure Prophylaxis
Keywords: PrEP; Community Health Worker; Criminal Justice
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: There will be two groups that participants can be assigned to if they choose to participate in the study. Each person will be randomly assigned to one of these groups. One group will provide information about PrEP and HIV prevention and referral to PrEP clinics in the community. The second group will the same as the first group but will also provide access to a CHW who will assist them with getting to a PrEP clinic and also helping them with other needs they may have.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Standard of Care (Active Comparator): PrEP education and referral to a community-based PrEP provider (enhanced standard of care)
  Interventions: Other: Enhanced Standard of Care
- Community Health Worker Involved Enhanced Standard of Care (Experimental): PrEP education, referral to a community-based PrEP provider, and referral to a CHW who will facilitate access to community-based PrEP and other healthcare and social-support services.
  Interventions: Behavioral: PrEP-LINK

INTERVENTIONS:
Behavioral: PrEP-LINK — CHW will assist with healthcare and social service navigation and will utilize adherence counseling techniques. As per the model our intervention is based upon (the national Transitions Clinic Network [TCN]), our CHW has a history of incarceration. Participants randomized to the intervention group, the CHW will assist individuals with employment, housing (if needed), referrals to mental health or substance use treatment, keeping track of medical appointments and medication adherence.
  Arms: Community Health Worker Involved Enhanced Standard of Care
Other: Enhanced Standard of Care — Participants will receive education about PrEP and referral to a community PrEP provider which exceeds the standards of care these individuals would otherwise receive.
  Arms: Enhanced Standard of Care

SUMMARY:
Our proposed study will: provide a novel exploration of facilitators and barriers to PrEP; allow us to target hard to reach populations, including men who have sex with men (MSM) and substance users (both of which are top funding priority groups for the National Institutes of Health) who experience intersecting markers of HIV risk; and inform regional, and possibly national, intervention approaches to combat the overlapping epidemic of HIV and incarceration.

DETAILED DESCRIPTION:
Specific Aims

The specific aims of the project associated with this protocol are:

Aim 1: Perform a qualitative assessment of facilitators and barriers to PrEP uptake among high-risk jail detainees, systems and interactor levels. To achieve this aim we will conduct qualitative interviews with three distinct groups of stakeholders:

1. Systems interviews (n=6);
2. Interactor interviews (n=8); and
3. Individual Key Informant interviews (n=20).

Within each of these strata, we aim to collect data representing diverse perspectives with respect to interest, knowledge, attitudes, and barriers (including substance use) to PrEP uptake. We will also explore acceptability and feasibility of an intervention to link individuals being released from the Pulaski County jail to PrEP services.

For the purposes of this protocol, Aims 2 and 3 are identical in terms of participant recruitment, enrollment and all study procedures (including data collection and participant follow up). The primary objective of Aim 2 is to conduct a small pilot of the intervention study in order to make any necessary changes to any aspect of the study procedures. If any changes are made, those changes will be submitted to the IRB for further review and approval prior to initiating Aim 3. If no changes are made, this IRB protocol will serve as the protocol for both Aims 2 and 3.

Aim 2: Develop the PrEP-LINK intervention and perform an open label evaluation with high-risk HIV negative individuals being discharged from the Pulaski County Jail or recently discharged from a correctional setting and reporting to a local Community Corrections facility or Re-Entry Center, including: Central Arkansas Community Corrections Center, East Central Arkansas Community Corrections Center, Hidden Creek Opportunity Center, Quality Living Center, Better Community Development, Inc., and Recovery Centers of Arkansas, .Directly informed from formative work (Aim 1), we will develop the PrEP-LINK intervention, which will include the use of a community health worker (CHW) and adherence counseling (based on ADAPT-ITT) approach to enhance PrEP care and overcome barriers to uptake in this population. We will then perform an open pilot with individuals recently released from a correctional facility

Aim 3: Conduct a pilot RCT of the PrEP-LINK intervention among high-risk HIV negative individuals being released from the Pulaski County Jail or recruited within 30 days of release from a correctional facility. Based on the formative work in Aim 1 and open pilot evaluation in Aim 2, participants will be randomized to either the PrEP-LINK intervention, or enhanced standard of care arm. Both arms will receive education about PrEP and referral to a community PrEP provider which exceeds the standards of care these individuals would otherwise receive.

While we will develop the CHW intervention as part of Aim 2, this will be informed by work we have already completed through Aim 1, which was approved under a separate IRB protocol (#207297). Once we have finalized the intervention content, we will conduct the Aim 2 open label evaluation in the exact same way as we will conduct the Aim 3 pilot RCT. To reiterate, the rationale of the open label evaluation proposed in Aim 2 is to ensure that the intervention is appropriate and does not need additional revision prior to conducting the Aim 3 RCT.

Description of the Community Health Worker (CHW) Intervention (Aims 2 and 3): The intervention arm in both Aims 2 and 3 will receive additional support by a community health worker (CHW) who will assist with healthcare and social service navigation and will utilize adherence counseling techniques. The CHW we are employing is Ms. Timikia Jackson, who is a trained CHW with a strong knowledge base of both healthcare and social service systems in the greater Little Rock area. As per the model our intervention is based upon (the national Transitions Clinic Network [TCN], which has 14 sites across the country), Ms. Jackson has a history of incarceration. Therefore, she can serve as a true peer to individuals who are enrolled into the study. The national TCN sites employ formerly incarcerated CHWs because these individuals are often able to develop close relationships with their peers who have also been formerly incarcerated thereby building a strong foundation of trust among a population with high levels of distrust of the medical system. Ms. Jackson will be certified in HIV testing and risk reduction counseling. For participants randomized to the intervention group, Ms. Jackson will assist individuals with employment, housing (if needed), referrals to mental health or substance use treatment, keeping track of medical appointments and medication adherence. We anticipate that Ms. Jackson will be in contact with intervention arm participants at least once per week but the exact amount of contact for each participant will vary based on needs. Ms. Jackson will be available during regular business hours (Monday-Friday, 9 AM until 5 PM). If participants present to Ms. Jackson in crisis, she will refer them immediately to the Emergency Department, in the event of a medical or behavioral health emergency or the Pulaski County Regional Crisis Stabilization Center, which is operated by the UAMS Psychiatric Research Institute (PRI). Ms.Jackson will be directly supervised by PI Dr. Zaller through weekly supervision meetings and biweekly phone check-ins. Frequency of check-in may increase or decrease, as needed, during the course of the study period. Ms. Jackson is considered research staff and has been trained in human subjects through the UAMS CITI program.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 at study enrollment
2. Able to understand and speak English and to provide written and verbal informed consent.
3. Able to provide reliable pieces of locator information (e.g. mailing address, phone number, email address, places frequently visited, etc.)
4. HIV negative confirmed through an on-site rapid HIV test;
5. Recently released from the Pulaski County Regional Detention Facility into the community and not into another detention facility or recently released (within 30 days) from a correctional facility and residing in Central Arkansas.
6. At substantial risk for HIV as determined by CDC/WHO PrEP guidelines, which includes engaging in any of the following behaviors in the last six months:

   * Having condomless vaginal or anal sex with more than one partner,
   * Having a sex partner with one or more HIV risk (e.g. PWID, a sex worker),
   * Being diagnosed with a STI,
   * Reporting history of sharing injection material/equipment, or
   * Having a sexual partner who is HIV positive.

Exclusion Criteria:

* Potential participants unable to provide informed consent, including people with severe mental illness requiring immediate treatment or with mental illness limiting their ability to participate (e.g., dementia), will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nickolas D Zaller, Ph.D, Principal Investigator — University of Arkansas
Locations (7):
- United States (7):
  - Better Community Development, Inc, Little Rock, Arkansas
  - Central Arkansas Community Corrections Center, Little Rock, Arkansas
  - Pulaski County County Regional Detention Facility, Little Rock, Arkansas
  - Quality Living Center, Little Rock, Arkansas
  - Recovery Centers of Arkansas, Little Rock, Arkansas
  - Hidden Creek Opportunity Center, Little Rock, Arkansas
  - East Central Arkansas Community Correction Center, West Memphis, Arkansas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enhanced Standard of Care | Community Health Worker Involved Enhanced Standard of Care
Started | 50 | 50
6 Month Assessment (6 month assessment completed.) | 19 | 20
Completed (12 month assessment completed.) | 20 | 16
Not Completed | 30 | 34
Not completed — Lost to Follow-up | 23 | 22
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Reincarcerated | 7 | 10
Not completed — Moved out of U.S. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Standard of Care | Community Health Worker Involved Enhanced Standard of Care | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.14 (8.65) | 37 (10.18) | 36.46 (9.49)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 29 | 27 | 56
  Female | 21 | 23 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 45 | 47 | 92
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 18 | 36
  White | 28 | 29 | 57
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction of the Utilization of the CHW to Aid in Accessing PrEP Assessed by the Client Satisfaction Questionnaire-Revised
Description: The acceptability of the intervention will be determined with descriptive statistics of the participants' acceptability ratings, including whether they think the intervention is acceptable. Acceptability is defined as > 80% of participants expressing high satisfaction with the intervention based on the Client Satisfaction Questionnaire - Revised (CSQ-8). The CSQ-8 is scored using a scale which ranges from 8-32, with a higher number indicating greater satisfaction.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score on CSQ-8
Arm/Group | Community Health Worker Involved Enhanced Standard of Care
Number analyzed (Participants) | 16
Score on CSQ-8 | 29.5 (3.26)

2. Primary Outcome: Rate of PrEP Uptake Among Participants Based on Medical Chart Review
Description: The preliminary efficacy of the intervention will be determined by assessing the primary outcome of PrEP uptake by looking at the medical charts of the participants. A secondary outcome will be PrEP adherence defined by participants who were adherent to the medication determined by self-report at 6, and 12 months.
Time Frame: 12 months
Population: No participants in either group reported taking PrEP at 12 month assessment, therefore medical chart review was not completed on any participant.
Arm/Group | Enhanced Standard of Care | Community Health Worker Involved Enhanced Standard of Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Rate of PrEP Adherence and Retention Based on Self-reported Surveys (PrEP-Use, PrEP-Attitude, PrEP-Adherence)
Description: A secondary outcome will be PrEP adherence defined by participants who were adherent to the medication determined by self-report at 6, and 12 months.
Time Frame: 6 months
Population: One participant in the Community Health Worker Involved Enhanced Standard of Care (intervention) arm reported currently taking PrEP at 6 month assessment (20 intervention arm participants completed the 6 month assessment). No participants in the Enhanced Standard of Care (control) arm reported currently taking PrEP at 6 month reassessment (18 control arm participants completed the 6 month assessment).
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Standard of Care | Community Health Worker Involved Enhanced Standard of Care
Number analyzed (Participants) | 18 | 20
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: This research was monitored for adverse events throughout the 12 month intervention (intervention arm only), and during the 6 month and 12 month follow-up assessments for both arms.
Arm/Group | Enhanced Standard of Care | Community Health Worker Involved Enhanced Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic forced closure of research activities within the original study recruitment site, the county detention center. The study team then shifted recruitment to community based re-entry settings. Barriers caused by the COVID-19 pandemic, conditions specific to re-entry centers, and competing priorities of those leaving incarceration may have all contributed to lack of study engagement and PrEP use. Some participants were reincarcerated within their year of study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT04064567/Prot_SAP_001.pdf